CLINICAL TRIAL: NCT06316401
Title: Endoscopic Submucosal Dissection of Large Recto-sigmoid Lesions Under Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Dr. Mauro Manno, Directore Gastroenterology and Endoscopy Unit, Azienda USL Modena
Other Study IDs: 03-2024
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Colorectal (Colon or Rectal) Cancer
Keywords: ESD; Spinal Anesthesia; colorectal lesions; LST; Laterally Spreading Tumor; endoscopic submucosal dissection; deep sedation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent endoscopic submucosal dissection under spinal anesthesia: We collected data on all consecutive patients who underwent ESD for recto-sigmoid laterally spreading tumors (LSTs) >35 mm under SA.
  SA was carried out in a sitting position, following a strictly aseptic technique. After recognition of L2-L3 intervertebral space through landmark technique, a 25 Gauge needle was inserted and the correct positioning was confirmed by detecting free flow of cerebrospinal fluid. Subsequently, 10-12 mg of hyperbaric bupivacaine + sufentanil 2 mcg according to the decision of the anesthetist was administered intrathecally without barbotage.
  Subsequently, the patient underwent ESD of the colorectal lesion.
  Interventions: Procedure: ESD of large LSTs under SA

INTERVENTIONS:
Procedure: ESD of large LSTs under SA — endoscopic submucosal dissection of large colorectal lesions under spinal anesthesia

SUMMARY:
The investigators collected data on all consecutive patients who underwent ESD for recto-sigmoid laterally spreading tumors (LSTs) >35 mm under SA between January 2021 and March 2024. The investigators evaluated the technical success and safety of SA in terms of ARAEs, and pain, measured via visual assessment scale (VAS).

DETAILED DESCRIPTION:
Background and study aim: Endoscopic submucosal dissection (ESD) of large colorectal lesions requires the patient to be in a still position for a long time. Both deep sedation and general anesthesia carry a substantial risk of anesthesia-related adverse events (ARAEs), especially in frail patients. Conversely, mild-to-moderate sedation does not prevent involuntary movements of the patient. Spinal anesthesia (SA) is a safe and simple technique that provides analgesia and motor block without systemic drug administration or orotracheal intubation. As the use of SA in colorectal endoscopic resections has not been described so far, we aimed to evaluate the feasibility and performance of SA in large (>35 mm) recto-sigmoid lesion ESD.

Patients and methods: The investigators collected data on all consecutive patients who underwent ESD for recto-sigmoid laterally spreading tumors (LSTs) >35 mm under SA between January 2021 and March 2024. The investigators evaluated the technical success and safety of SA in terms of ARAEs, and pain, measured via visual assessment scale (VAS). The secondary endpoints were as follows: intra- and post-procedural need for additional opioid or other analgesic drug administration, ESD-related adverse eventss, length of hospital stay, and median ESD duration.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* American Society of Anaesthesiologists (ASA) score I-IV
* ability to give informed consent

Exclusion Criteria:

* age <18 years
* ASA score V
* allergy to medications used for spinal anesthesia
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients eligibility underwent ESD for large LSTs under SA
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Technical success of ESD under SA | Immediately after the procedure
  Technical success was defined as completion of the ESD under SA without the need of conversion to deep sedation or general anesthesia.
Safety of ESD under SA | periprocedurally
  Safety was evaluated intra- and post-procedurally by recording anesthesia-related adverse events (ARAEs). Major ARAEs included death, anaphylaxis and severe cardiorespiratory or neurologic AEs. Minor ARAEs included any other cardiorespiratory or neurologic AEs, headache, acute urinary retention and itching.

SECONDARY OUTCOMES:
Intra- and post-procedural need for additional opioid or other analgesic drug administration | periprocedurally
  Intra- and post-procedural need for additional opioid or other analgesic drug administration
ESD- and colonoscopy-related AEs | periprocedurally
  Perforation, bleeding, post-coagulation syndrome, adverse events related to endoscopic bowel preparation
Length of hospital stay | At delivery
  length of hospital stay
Median ESD duration | Immediately after the procedure
  Median ESD duration

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manno, MD, Principal Investigator — AUSL Modena
Locations (1):
- Mauro Manno, Carpi, MO, Italy

IPD SHARING:
Plan to Share IPD: Undecided